CLINICAL TRIAL: NCT03496909
Title: The PhysioTouch, A Novel Treatment for Radiation Fibrosis Syndrome in Breast Cancer Patients
Brief Title: PhysioTouch for Treatment of Radiation Fibrosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Reduction in available resources
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Katie Rogers, Occupational Therapist, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00130272
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Radiation Fibrosis
MeSH Terms: conditions — Radiation Fibrosis Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard OT (Active Comparator)
  Interventions: Behavioral: Standard OT
- PhysioTouch (Experimental)
  Interventions: Behavioral: PhysioTouch

INTERVENTIONS:
Behavioral: Standard OT — 12 weekly sessions of occupational therapy tailored to patients with RFS secondary to breast cancer treatment. Sessions can include manual therapy, education, and active and passive range-of-motion, etc.
  Arms: Standard OT
Behavioral: PhysioTouch — 12 weekly sessions of occupational therapy tailored to patients with RFS secondary to breast cancer treatment. Sessions can include use of the PhysioTouch electronic massager in lieu of manual therapy, education, and active and passive range-of-motion, etc.
  Arms: PhysioTouch

SUMMARY:
A quarter of a million women will develop breast cancer (BC) in this year alone. Many of these women will have side effects as a result of their breast cancer treatment. Radiation Fibrosis Syndrome (RFS) is a common complication from breast cancer treatment that progressively changes tissue and can cause decreased function, pain, and range of motion. The PhysioTouch is a hand held device that can be used to treat RFS and may improve the treatment of fibrotic tissue. This pilot randomized controlled trial aims to determine the efficacy of using the PhysioTouch in addition to current standard of care for treatment of BC-related RFS.

ELIGIBILITY:
Inclusion Criteria:

* History of radiation therapy for breast cancer
* Clinical or suspected RFS
* Reported functional impairments

Exclusion Criteria:

* Metastatic disease of soft tissue
* History of bilateral radiation therapy
* Previously diagnosed shoulder impairments not related to RFS
* Prior treatment with PhysioTouch
* Current or recent pregnancy
* Current breastfeeding
* Other contraindications to safe and meaningful participation at discretion of study team

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported upper extremity function | Baseline to 12 weeks
  Self-reported upper extremity function as measured by QuickDash
Change in self-reported pain | Baseline to 12 weeks
  Self-reported upper extremity pain as measured by the BPI

SECONDARY OUTCOMES:
Change in affected shoulder abduction | Baseline to 12 weeks
  Degrees of should abduction as measured by OT
Change in affected shoulder flexion | Baseline to 12 weeks
  Degrees of should flexsion as measured by OT

CONTACTS AND LOCATIONS:
Overall Officials: Katie Rogers, MSOTR-CLT, Principal Investigator — Michigan Medicine, Department of Physical Medicine & Rehabiliation